CLINICAL TRIAL: NCT00952289
Title: A Randomized, Double-blind, Placebo-controlled Study of the JAK Inhibitor INCB018424 Tablets Administered Orally to Subjects With Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis or Post-Essential Thrombocythemia Myelofibrosis
Brief Title: COntrolled MyeloFibrosis Study With ORal JAK Inhibitor Treatment: The COMFORT-I Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 18424-351
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2012-01-24 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: MPN (Myeloproliferative Neoplasms)
Keywords: Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ruxolitinib (Experimental): Participants received ruxolitinib orally twice a day. The starting dose was determined based on Baseline platelet count. Patients with Baseline platelet count > 200,000/μL began a dose regimen of 20 mg twice daily. Patients with Baseline platelet count of 100,000/μL to 200,000/μL (inclusive) began a dose regimen of 15 mg twice daily. The dose was adjusted by the Investigator based on efficacy and safety to a maximum of 25 mg twice daily. Patients receiving benefit could continue treatment until the later of marketing approval or when the last randomized patient remaining in the study had completed Week 144 (36 months).
  Interventions: Drug: Ruxolitinib
- Placebo (Placebo Comparator): Placebo tablets matching ruxolitinib were administered orally twice a day at a starting dose based on Baseline platelet count. Doses were titrated using the same guidelines as for active drug. Patients meeting certain protocol requirements detailed below were given the opportunity to cross over to ruxolitinib treatment.
  Interventions: Drug: Ruxolitinib; Drug: Placebo

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib phosphate tablets 5 mg administered as oral doses.
  Other Names: INCB018424
Drug: Placebo — Matching placebo tablets were administered as oral doses in the same manner as active drug.
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind study comparing the efficacy and safety of ruxolitinib (INCB018424) tablets to matching placebo tablets in patients diagnosed with Myelofibrosis (either Primary Myelofibrosis (PMF) or Post-Polycythemia Vera Myelofibrosis (PPV-MF) or Post-Essential Thrombocythemia Myelofibrosis (PET-MF).

DETAILED DESCRIPTION:
Patients with spleen growth of greater than 25% based on an increase in spleen volume from Baseline were eligible for early unblinding, and for patients on placebo, cross over to ruxolitinib prior to the primary study endpoint being reached. If this spleen growth occurred before Week 24, it must have been accompanied by specific worsening of symptoms, based on worsening early satiety accompanied by weight loss or worsening pain requiring daily narcotic use. After Week 24, asymptomatic spleen growth alone was sufficient for early unblinding and potential cross over. Patients found to have been randomized to ruxolitinib after early unblinding prior to Week 24 were discontinued.

When half of the patients remaining in the study completed the Week 36 visit and all patients enrolled completed Week 24 or discontinued, the database was frozen and the primary analysis was conducted. Once this was complete, all patients were unblinded and patients who had been randomized to placebo were given the opportunity to cross over to ruxolitinib treatment, provided hematology laboratory parameters were adequate; Patients receiving benefit could continue treatment until the later of marketing approval or when the last randomized patient remaining in the study had completed Week 144 (36 months).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be diagnosed with primary myelofibrosis (PMF), post-polycythemia vera-myelofibrosis (PPV-MF) or post-essential thrombocythemia-myelofibrosis (PET-MF) according to the 2008 World Health Organization criteria
* Subjects with myelofibrosis requiring therapy must be classified as high risk OR intermediate risk level 2 according to the prognostic factors defined by the International Working Group
* Subjects with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2 or 3
* Subjects who have not previously received treatment with a Janus kinase (JAK) inhibitor

Exclusion Criteria:

* Subjects with a life expectancy of less than 6 months
* Subjects with inadequate bone marrow reserve as demonstrated by specific clinical laboratory counts
* Subjects with inadequate liver or renal function
* Subjects with clinically significant bacterial, fungal, parasitic or viral infection which require therapy
* Subjects with an active malignancy over the previous 5 years except specific skin cancers.
* Subjects with severe cardiac conditions
* Subjects who have had splenic irradiation within 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, MD, PhD, Study Director — M.D. Anderson Cancer Center
Locations (112):
- United States (88):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Baldwin Park, California
  - Bellflower, California
  - Beverly Hills, California
  - Corona, California
  - Fullerton, California
  - Highland, California
  - La Jolla, California
  - Los Angeles, California
  - Orange, California
  - Palo Alto, California
  - Panorama City, California
  - Rancho Cucamonga, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - West Covina, California
  - Aurora, Colorado
  - Denver, Colorado
  - Fort Collins, Colorado
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Boynton Beach, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Honolulu, Hawaii
  - Boise, Idaho
  - Meridian, Idaho
  - Twin Falls, Idaho
  - Chicago, Illinois
  - Beech Grove, Indiana
  - Indianapolis, Indiana
  - Ames, Iowa
  - Iowa City, Iowa
  - Sioux City, Iowa
  - Waterloo, Iowa
  - Louisville, Kentucky
  - Alexandria, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Novi, Michigan
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Saint Louis Park, Minnesota
  - New Albany, Mississippi
  - St Louis, Missouri
  - Billings, Montana
  - Denville, New Jersey
  - Hackensack, New Jersey
  - Morristown, New Jersey
  - Somerville, New Jersey
  - Albuquerque, New Mexico
  - East Setauket, New York
  - New York, New York
  - Valhalla, New York
  - Durham, North Carolina
  - Hickory, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Akron, Ohio
  - Canton, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Dover, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Germantown, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - New Braunfels, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Everett, Washington
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Australia (16):
  - Darlinghurst, New South Wales
  - Kogarah, New South Wales
  - Randwick, New South Wales
  - St Leonards, New South Wales
  - Brisbane, Queensland
  - Douglas, Queensland
  - Herston, Queensland
  - Milton, Queensland
  - Woolloongabba, Queensland
  - Bedford Park, South Australia
  - Box Hill, Victoria
  - Clayton, Victoria
  - Frankston, Victoria
  - Ringwood East, Victoria
  - Fremantle, Western Australia
  - Perth, Western Australia
- Canada (8):
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Lévis, Quebec
  - Montreal, Quebec

REFERENCES:
- [Background] Verstovsek S, Mesa R, Gotlib J, et al. Results of COMFORT-I, a randomized double-blind phase III trial of JAK1/2 inhibitor INCB18424 (424) vs placebo (PB) for patients with myelofibrosis (MF). The 47th Annual ASCO meeting, Chicago, IL. J Clin Oncol 2011; 29 (suppl; abstract 6500). Verstovsek S, Mesa R, Gotlib J, et al. Results of COMFORT-I, a randomized, double-blind phase III trial of the JAK1 and JAK2 inhibitor ruxolitinib (INCB018424) versus placebo for patients with myelofibrosis. The 16th Annual EHA meeting, London, UK. Haematologica 2011; 96 (suppl 2; abstract 0505).
- [Result] Verstovsek S, Mesa RA, Gotlib J, Levy RS, Gupta V, DiPersio JF, Catalano JV, Deininger M, Miller C, Silver RT, Talpaz M, Winton EF, Harvey JH Jr, Arcasoy MO, Hexner E, Lyons RM, Paquette R, Raza A, Vaddi K, Erickson-Viitanen S, Koumenis IL, Sun W, Sandor V, Kantarjian HM. A double-blind, placebo-controlled trial of ruxolitinib for myelofibrosis. N Engl J Med. 2012 Mar 1;366(9):799-807. doi: 10.1056/NEJMoa1110557. PMID 22375971
- [Result] Verstovsek S, Mesa RA, Gotlib J, Levy RS, Gupta V, DiPersio JF, Catalano JV, Deininger MW, Miller CB, Silver RT, Talpaz M, Winton EF, Harvey JH Jr, Arcasoy MO, Hexner EO, Lyons RM, Paquette R, Raza A, Vaddi K, Erickson-Viitanen S, Sun W, Sandor V, Kantarjian HM. Efficacy, safety and survival with ruxolitinib in patients with myelofibrosis: results of a median 2-year follow-up of COMFORT-I. Haematologica. 2013 Dec;98(12):1865-71. doi: 10.3324/haematol.2013.092155. Epub 2013 Sep 13. PMID 24038026
- [Result] Verstovsek S, Mesa RA, Gotlib J, Levy RS, Gupta V, DiPersio JF, Catalano JV, Deininger MW, Miller CB, Silver RT, Talpaz M, Winton EF, Harvey JH Jr, Arcasoy MO, Hexner EO, Lyons RM, Raza A, Vaddi K, Sun W, Peng W, Sandor V, Kantarjian H; COMFORT-I investigators. Efficacy, safety, and survival with ruxolitinib in patients with myelofibrosis: results of a median 3-year follow-up of COMFORT-I. Haematologica. 2015 Apr;100(4):479-88. doi: 10.3324/haematol.2014.115840. Epub 2015 Jan 23. PMID 25616577
- [Derived] Verstovsek S, Gotlib J, Mesa RA, Vannucchi AM, Kiladjian JJ, Cervantes F, Harrison CN, Paquette R, Sun W, Naim A, Langmuir P, Dong T, Gopalakrishna P, Gupta V. Long-term survival in patients treated with ruxolitinib for myelofibrosis: COMFORT-I and -II pooled analyses. J Hematol Oncol. 2017 Sep 29;10(1):156. doi: 10.1186/s13045-017-0527-7. PMID 28962635
- [Derived] Miller CB, Komrokji RS, Mesa RA, Sun W, Montgomery M, Verstovsek S. Practical Measures of Clinical Benefit With Ruxolitinib Therapy: An Exploratory Analysis of COMFORT-I. Clin Lymphoma Myeloma Leuk. 2017 Aug;17(8):479-487. doi: 10.1016/j.clml.2017.05.015. Epub 2017 May 12. PMID 28606598
- [Derived] Verstovsek S, Mesa RA, Gotlib J, Gupta V, DiPersio JF, Catalano JV, Deininger MW, Miller CB, Silver RT, Talpaz M, Winton EF, Harvey JH Jr, Arcasoy MO, Hexner EO, Lyons RM, Paquette R, Raza A, Jones M, Kornacki D, Sun K, Kantarjian H; COMFORT-I investigators. Long-term treatment with ruxolitinib for patients with myelofibrosis: 5-year update from the randomized, double-blind, placebo-controlled, phase 3 COMFORT-I trial. J Hematol Oncol. 2017 Feb 22;10(1):55. doi: 10.1186/s13045-017-0417-z. PMID 28228106
- [Derived] Deininger M, Radich J, Burn TC, Huber R, Paranagama D, Verstovsek S. The effect of long-term ruxolitinib treatment on JAK2p.V617F allele burden in patients with myelofibrosis. Blood. 2015 Sep 24;126(13):1551-4. doi: 10.1182/blood-2015-03-635235. Epub 2015 Jul 30. PMID 26228487
- [Derived] Vannucchi AM, Kantarjian HM, Kiladjian JJ, Gotlib J, Cervantes F, Mesa RA, Sarlis NJ, Peng W, Sandor V, Gopalakrishna P, Hmissi A, Stalbovskaya V, Gupta V, Harrison C, Verstovsek S; COMFORT Investigators. A pooled analysis of overall survival in COMFORT-I and COMFORT-II, 2 randomized phase III trials of ruxolitinib for the treatment of myelofibrosis. Haematologica. 2015 Sep;100(9):1139-45. doi: 10.3324/haematol.2014.119545. Epub 2015 Jun 11. PMID 26069290
- [Derived] Mesa RA, Verstovsek S, Gupta V, Mascarenhas JO, Atallah E, Burn T, Sun W, Sandor V, Gotlib J. Effects of ruxolitinib treatment on metabolic and nutritional parameters in patients with myelofibrosis from COMFORT-I. Clin Lymphoma Myeloma Leuk. 2015 Apr;15(4):214-221.e1. doi: 10.1016/j.clml.2014.12.008. Epub 2014 Dec 27. PMID 25682576
- [Derived] Mesa RA, Kiladjian JJ, Verstovsek S, Al-Ali HK, Gotlib J, Gisslinger H, Levy R, Siulnik A, Gupta V, Khan M, DiPersio JF, McQuitty M, Catalano JV, Hunter DS, Knoops L, Deininger M, Cervantes F, Miller C, Vannucchi AM, Silver RT, Barbui T, Talpaz M, Barosi G, Winton EF, Mendeson E, Harvey JH Jr, Arcasoy MO, Hexner E, Lyons RM, Paquette R, Raza A, Sun W, Sandor V, Kantarjian HM, Harrison C. Comparison of placebo and best available therapy for the treatment of myelofibrosis in the phase 3 COMFORT studies. Haematologica. 2014 Feb;99(2):292-8. doi: 10.3324/haematol.2013.087650. Epub 2013 Aug 2. PMID 23911705
- [Derived] Mesa RA, Gotlib J, Gupta V, Catalano JV, Deininger MW, Shields AL, Miller CB, Silver RT, Talpaz M, Winton EF, Harvey JH, Hare T, Erickson-Viitanen S, Sun W, Sandor V, Levy RS, Kantarjian HM, Verstovsek S. Effect of ruxolitinib therapy on myelofibrosis-related symptoms and other patient-reported outcomes in COMFORT-I: a randomized, double-blind, placebo-controlled trial. J Clin Oncol. 2013 Apr 1;31(10):1285-92. doi: 10.1200/JCO.2012.44.4489. Epub 2013 Feb 19. PMID 23423753

RESULTS

PARTICIPANT FLOW:
Groups:
- Ruxolitinib: Participants received ruxolitinib orally twice a day. The starting dose was based on Baseline platelet count. Patients with Baseline platelet count > 200,000/μL began a dose regimen of 20 mg twice daily. Patients with Baseline platelet count of 100,000/μL to 200,000/μL (inclusive) began a dose regimen of 15 mg twice daily. The dose was adjusted by the Investigator based on efficacy and safety to a maximum of 25 mg twice daily. Patients receiving benefit could continue treatment until the later of marketing approval or when the last randomized patient remaining in the study had completed Week 144 (36 months).
- Placebo: Placebo tablets matching ruxolitinib were administered orally twice a day at a starting dose based on Baseline platelet count. Doses were titrated using the same guidelines as for active drug. Patients meeting pre-specified requirements were given the opportunity to cross over to ruxolitinib treatment.
Period: All Participants
Arm/Group | Ruxolitinib | Placebo
Started | 155 | 154
Safety Population | 155 | 151 (Randomized patients who are documented to have received at least 1 dose of study medication.)
Completed | 134 (Represents the number of patients who were still in the study as of 02 November 2010) | 114 (Includes patients in the study as of 2 November 2010 (78) + those who crossed over to Ruxolitinib.)
Not Completed | 21 | 40
Not completed — Death | 9 | 9
Not completed — Adverse Event | 8 | 8
Not completed — Disease progression | 3 | 12
Not completed — Withdrawal by Subject | 1 | 10
Not completed — Data lost during site relocation | 0 | 1
Period: Patients Who Crossed Over to Ruxolitinib
Arm/Group | Ruxolitinib | Placebo
Started | 0 | 111
Completed | 0 | 57 (Number of cross over subjects who were still in the study as of 25 JAN 2013)
Not Completed | 0 | 54
Not completed — Adverse Event | 0 | 19
Not completed — Disease progression | 0 | 15
Not completed — Withdrawal by Subject | 0 | 11
Not completed — Non-compliance to study medication | 0 | 2
Not completed — Other Unspecified | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Ruxolitinib: Participants began treatment with ruxolitinib 15 or 20 mg taken orally twice a day based on Baseline platelet count. The dose was adjusted by the Investigator based on efficacy and safety to a maximum of 25 mg twice daily.
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib | Placebo | Total
Number analyzed (Participants) | 155 | 154 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.7 (8.82) | 68.7 (8.66) | 67.7 (8.78)
Sex/Gender, Customized [Number; unit: participants] — Population: Gender data for one patient in the placebo arm was not available because of loss of study data during a move to a new location by the clinical site.
  participants
    Female: number analyzed (Participants) | 155 | 153 | 308
    Female | 76 | 65 | 141
    Male: number analyzed (Participants) | 155 | 153 | 308
    Male | 79 | 88 | 167
Race/Ethnicity, Customized [Number; unit: participants] — Race data for one patient in the placebo arm was not available because of loss of study data during a move to a new location by the clinical site.
  participants
    Black or African American | 6 | 7 | 13
    White | 138 | 139 | 277
    Asian | 5 | 4 | 9
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Other | 5 | 3 | 8
Disease Subtype [Number; unit: participants]
  Primary myelofibrosis | 70 | 84 | 154
  Post-polycythemia vera-myelofibrosis | 50 | 47 | 97
  Post-essential thrombocythemia-myelofibrosis | 35 | 22 | 57
  Missing | 0 | 1 | 1
Spleen volume [Mean (Standard Deviation); unit: cm˄3] — Spleen volume was measured by magnetic resonance imaging or computed tomography scans. Data for one patient in the placebo arm was not available because of loss of study data during a move by the clinical site.
  cm˄3 | 2745.7 (1247.0) | 2797.6 (1388.5) | 2771.5 (1317.3)
JAK2 V617F Mutation Status [Number; unit: participants] — JAK2V617F is a mutation in the pseudokinase domain of Janus Kinase 2 (JAK2) (at amino acid 617, valine to phenylalanine) that results in constitutive activation of JAK2. Mutation status was determined using a validated assay on bone marrow as well as peripheral blood.
  participants
    Positive | 113 | 123 | 236
    Negative | 40 | 27 | 67
    Unknown/Missing | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving ≥ 35% Reduction in Spleen Volume From Baseline to Week 24
Description: Spleen volume was assessed by magnetic resonance imaging (MRI) or by computed tomography (CT) scans if MRI was not suitable, and analyzed by a blinded central laboratory reader. Patients who withdrew, crossed over to ruxolitinib prior to the visit, or had a missing value at the visit were considered non-responders.
Time Frame: Baseline and Week 24
Population: Intent-to-treat (ITT) population included all subjects randomized in the study. Treatment groups for this population were defined according to the treatment assignment at randomization. One patient was not included in the analysis due to a missing baseline spleen volume value.
Measure: Number; unit: participants
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 155 | 153
participants | 65 | 1
Statistical Analysis 1: Comparison: Ruxolitinib vs Placebo; The primary endpoint analyzed with a 2-sided alpha of 0.05; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Secondary Outcome: Maintenance of a ≥ 35% Reduction From Baseline in Spleen Volume Among Patients Initially Randomized to Receive Ruxolitinib
Description: The maintenance of ≥ 35% reduction from Baseline in spleen volume was assessed up until the data cutoff date using the Kaplan-Meier method for patients who had at least one measured ≥ 35% reduction, and who either had at least one subsequent measurement or who subsequently dropped out prior to another assessment.
Time Frame: Baseline Visit and every 12 weeks until the data cut-off date (up to 14 months).
Population: Patients who had at least 1 measurement of ≥ 35% reduction from Baseline in spleen volume at any time during the study and had at least 1 subsequent measurement or withdrew prior to another assessment.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 91
proportion of participants
  Still Responder by 48 weeks | 0.76 [0.66 to 0.84]
  Still Responder by 96 weeks | 0.67 [0.55 to 0.76]
  Still Responder by 144 weeks | 0.27 [0.02 to 0.63]

3. Secondary Outcome: Duration of Maintenance of a ≥ 35% Reduction From Baseline in Spleen Volume Among Patients Initially Randomized to Receive Ruxolitinib
Description: The duration of ≥ 35% reduction from Baseline in spleen volume was defined as the longest duration of consecutive measurements of ≥ 35% reduction observed before the data cut-off date for patients who had at least one measured ≥ 35% reduction, and who either had at least one subsequent measurement or, who subsequently dropped out prior to another assessment. The duration of a ≥ 35% reduction from Baseline in spleen volume was analyzed using the Kaplan-Meier method.
Time Frame: Baseline Visit and every 12 weeks until the data cut-off date (up to 14 months).
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 91
weeks | 135.0 [107.6 to NA] — Data not evaluable due to a single loss of response with few subjects having spleen measurement follow-up data beyond 128 weeks from start of response.

4. Secondary Outcome: Number of Participants With a ≥ 50% Reduction in Total Symptom Score From Baseline to Week 24
Description: Symptoms of myelofibrosis were assessed using a modified Myelofibrosis Symptom Assessment Form (MFSAF) Version 2.0 diary. Using the diary, patients rated the following symptoms on a scale from 0 (absent) to 10 (worst imaginable): night sweats, itching, abdominal discomfort, pain under ribs on left, feeling of fullness (early satiety), and muscle/bone pain. The total symptom score ranged from 0-60 and was calculated as the sum of the 6 symptom scores. A higher score indicates worse symptoms.
Time Frame: Baseline and Week 24. Baseline total score was the average of the daily total scores for the last 7 days prior to randomization. The Week 24 total score was the average of daily total scores from the 28 days prior to the Week 24 visit.
Population: ITT evaluable population included patients with Baseline data and who did not have a 0 total score at both Baseline & Week 24; data measured after the cross over date were excluded. Patients who withdrew, met cross over criteria prior to Week 24 or had a 0 Baseline score & a nonzero/missing score at Week 24 were considered not meeting the endpoint.
Measure: Number; unit: participants
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 148 | 152
participants | 68 | 8

5. Secondary Outcome: Change From Baseline to Week 24 in Total Symptom Score
Description: Symptoms of myelofibrosis were assessed using a modified Myelofibrosis Symptom Assessment Form (MFSAF) Version 2.0 diary. Using the diary, patients rated the following symptoms on a scale from 0 (absent) to 10 (worst imaginable): night sweats, itching, abdominal discomfort, pain under ribs on left, feeling of fullness (early satiety), and muscle/bone pain. The total symptom score ranged from 0-60 and was calculated as the sum of the 6 symptom scores. A higher score indicates worse symptoms hence a negative change from baseline indicates improvement.
Time Frame: as for outcome 4
Population: This analysis only includes patients who had a non-missing change from Baseline to Week 24. Data collected after the date of treatment cross over were not included in this analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 131 | 105
scores on a scale
  Baseline | 18.0 (10.9) | 16.5 (11.5)
  Week 24 | 9.4 (9.7) | 19.7 (13.7)
  Change from Baseline | -8.6 (10.0) | 3.2 (9.4)

6. Secondary Outcome: Overall Survival
Description: Overall survival is reported here by the number of deaths from randomization until the data cut-off. Patients were censored at the time of database cut-off or the later of either the date of withdrawal or the date of last follow-up for patients who withdrew from study before the date of data cut. The survival time was analyzed using the Kaplan-Meier method.
Time Frame: From randomization to the data cut-off date (up to 14 months).
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 155 | 154
participants
  Death events | 10 | 14
  Censored events | 145 | 140

7. Secondary Outcome: Overall Survival Time
Description: Overall survival was assessed by the time to death or censoring. Patients were censored at the time of database cut-off or the later of either the date of withdrawal or the date of last follow-up for patients who withdrew from study before the date of data cut. The survival time was analyzed using the Kaplan-Meier method.
Time Frame: From randomization to the data cut-off date (up to 14 months).
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 155 | 154
weeks | NA [NA to NA] — The median overall survival was not reached as more than 50% of patients were still live at the time of the data cut-off using the Kaplan-Meier method. | NA [NA to NA] — The median overall survival was not reached as more than 50% of patients were still live at the time of the data cut-off using the Kaplan-Meier method.

8. Secondary Outcome: Overall Survival - Extended Data
Description: Overall survival is reported here by the number of deaths from randomization until 01 March 2011. Patients were censored at this time or the later of either the date of withdrawal or the date of last follow-up for patients who withdrew from study before the date of data cut. The survival time was analyzed using the Kaplan-Meier method. This outcome reports data from August 2009 through March 2011 to coincide with a pre-planned New Drug Application (NDA) 120-day safety update.
Time Frame: From randomization to 4 months after the data cut-off date (up to 18 months).
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 155 | 154
participants
  Death events | 13 | 24
  Censored events | 142 | 130

9. Secondary Outcome: Overall Survival Time - Extended Data
Description: Overall survival was assessed by the time to death or censoring up until 01 March 2011. Patients were censored at this time or the later of either the date of withdrawal or the date of last follow-up for patients who withdrew from study before the date of data cut. The survival time was analyzed using the Kaplan-Meier method. This outcome reports data from August 2009 through March 2011 to coincide with a pre-planned New Drug Application (NDA) 120-day safety update.
Time Frame: From randomization to 4 months after the data cut-off date (up to 18 months).
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 155 | 154
weeks | NA [NA to NA] — The median overall survival was not reached as more than 50% of patients were still living at the time of the database cut-off using the Kaplan-Meier method. | NA [NA to NA] — The median overall survival was not reached as more than 50% of patients were still living at the time of the database cut-off using the Kaplan-Meier method.

10. Secondary Outcome: Overall Survival at Week 144
Description: Overall survival is reported here by the number of deaths from randomization until the data cut-off. Patients were censored at the time of database cut-off or the later of either the date of withdrawal or the date of last follow-up for patients who withdrew from study before the date of database cut-off. The survival time was analyzed using the Kaplan-Meier method.
Time Frame: Week 144
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 155 | 154
participants
  Death events | 42 | 54
  Censored events | 113 | 100

11. Secondary Outcome: Overall Survival Time at Week 144
Description: Overall survival was assessed by the time to death or censoring. Patients were censored at the time of database cut-off or the later of either the date of withdrawal or the date of last follow-up for patients who withdrew from study before the date of database cut-off. The survival time was analyzed using the Kaplan-Meier method.
Time Frame: Week 144
Population: ITT population
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Ruxolitinib | Placebo
Number analyzed (Participants) | 155 | 154
probability | 0.74 [0.66 to 0.81] | 0.61 [0.53 to 0.69]

ADVERSE EVENTS:
Time Frame: From randomization through data cut-off of the primary analysis (02 November 2010).
Arm/Group | Ruxolitinib | Placebo
Serious Adverse Events (participants affected / at risk) | 43/155 | 53/151
Other Adverse Events (participants affected / at risk) | 150/155 | 147/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=155) | Placebo (N=151)
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 6
Ascites (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 1
Disease progression (General disorders) | 0 | 3
Fatigue (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 10 | 5
Sepsis (Infections and infestations) | 1 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Haemoglobin decreased (Investigations) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 3
Diverticulum (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Obturator hernia (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 1 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Splenic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Splenic injury (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Blast cells present (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (N=155) | Placebo (N=151)
Thrombocytopenia (Blood and lymphatic system disorders) | 52 | 14
Anaemia (Blood and lymphatic system disorders) | 45 | 20
Leukocytosis (Blood and lymphatic system disorders) | 1 | 8
Abdominal pain (Gastrointestinal disorders) | 16 | 58
Diarrhoea (Gastrointestinal disorders) | 36 | 32
Nausea (Gastrointestinal disorders) | 22 | 29
Constipation (Gastrointestinal disorders) | 20 | 18
Vomiting (Gastrointestinal disorders) | 18 | 15
Abdominal distension (Gastrointestinal disorders) | 13 | 16
Abdominal pain upper (Gastrointestinal disorders) | 9 | 13
Dyspepsia (Gastrointestinal disorders) | 9 | 8
Flatulence (Gastrointestinal disorders) | 8 | 1
Fatigue (General disorders) | 38 | 51
Oedema peripheral (General disorders) | 29 | 34
Pyrexia (General disorders) | 16 | 10
Asthenia (General disorders) | 6 | 12
Early satiety (General disorders) | 1 | 13
Pain (General disorders) | 4 | 9
Chills (General disorders) | 8 | 3
Performance status decreased (General disorders) | 2 | 9
Hepatomegaly (Hepatobiliary disorders) | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 9 | 13
Urinary tract infection (Infections and infestations) | 11 | 5
Nasopharyngitis (Infections and infestations) | 2 | 9
Haemoglobin decreased (Investigations) | 19 | 6
Platelet count decreased (Investigations) | 15 | 4
Cardiac murmur (Investigations) | 11 | 5
Blast cell count increased (Investigations) | 4 | 10
Weight increased (Investigations) | 10 | 2
Weight decreased (Investigations) | 0 | 9
Blood uric acid increased (Investigations) | 0 | 8
Anorexia (Metabolism and nutrition disorders) | 9 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Dizziness (Nervous system disorders) | 23 | 10
Headache (Nervous system disorders) | 23 | 8
Insomnia (Psychiatric disorders) | 18 | 15
Anxiety (Psychiatric disorders) | 3 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Rales (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Ecchymosis (Skin and subcutaneous tissue disorders) | 29 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 23
Night sweats (Skin and subcutaneous tissue disorders) | 10 | 18
Rash (Skin and subcutaneous tissue disorders) | 7 | 8
Erythema (Skin and subcutaneous tissue disorders) | 1 | 9
Pallor (Vascular disorders) | 8 | 9
Hypotension (Vascular disorders) | 5 | 8
Blood alkaline phosphatase increased (Investigations) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.